CLINICAL TRIAL: NCT02125968
Title: Therapeutic Effects of Video Game Play Therapy on Patients With Chronic Low Back Pain:Randomized-Controlled Clinical Trail
Brief Title: Therapeutic Effects of Video Game Play Therapy on Patients With Chronic Low Back Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKH-8302-103-DR-36
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; video game; therapeutic effects
MeSH Terms: interventions — Time; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- interactive video game (Active Comparator): Participants in interactive video game group receive six 20-min sessions of hot pack therapy combined 20-min of diathermy therapy over the low back followed by 15-min interactive video game intervention, for 3 times per week for a 2-week duration.
  Short- and medium-term therapeutic effects of interactive video game intervention for patients with chronic low back pain will be assessed.
  Interventions: Other: interactive video game
- therapeutic exercise (Sham Comparator): Participants received six 20-min sessions of hot pack therapy combined 20-min of diathermy therapy over the low back followed by 15-min supervised therapeutic exercise,for 3 times per week for a 2-week duration.
  short- and medium-term therapeutic effects of video game play therapy for patients with chronic low back pain will be evaluated.
  Interventions: Other: therapeutic exercise

INTERVENTIONS:
Other: interactive video game — short- and medium-term therapeutic effects
  Other Names: 6 sessions of 15-min, for a 2-week duration
  Arms: interactive video game
Other: therapeutic exercise — short- and medium-term therapeutic effects
  Other Names: 6 sessions of 15 min ,for a 2-week duration.
  Arms: therapeutic exercise

SUMMARY:
The purpose of this study is to investigate the video game play therapy in patients with chronic low back pain.

DETAILED DESCRIPTION:
Understanding the short- and medium-term therapeutic effects of video game play therapy for patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain

Exclusion Criteria:

1. low back pain accompanied by specific pathological conditions, such as infection, inflammation, fracture, or tumor
2. history of low back surgery with an implant
3. pregnancy of plans to become pregnant during the course of study
4. having received concurrent treatment for low back pain followed by another health care professional

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Questionnaire | changes from baseline at one and three months after treatment

SECONDARY OUTCOMES:
range of motion | changes from baseline at one and three months after treatment
Hospital Anxiety and Depression Scale | changes from baseline at one and three months after treatment
postural stability | changes from baseline at one and three months after treatment
  postural stability, limits of stability, and fall risk measured by Biodex Stability System
Fear avoidance Behavior Questionnaire | changes from baseline at one and three months after treatment
physical activity | changes from baseline at one and three months after treatment
  timed stairs climbing, 10-m walking, chair-rising time

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipie, Taiwan